CLINICAL TRIAL: NCT02328729
Title: Incident and Extent of Pulse Alteration During Administration of Various Modes of Local Anesthesia in Children During Routine Dental Treatment
Brief Title: Incident and Extent of Pulse Alteration During Local Anesthesia in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Sheba Medical Center (Other Government); Private practice, Dr. Malka Ashkenazi (Unknown)
Responsible Party: Principal Investigator, Mickey Scheinowitz, PhD, PhD, Tel Aviv University
Other Study IDs: 9995-12
Record Dates: First submitted 2014-12-25; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia | interventions — Epinephrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Mandibular block with Epinephrine: Lidocaine 2% with 1:100,000 Epinephrine
  Interventions: Procedure: mandibular block with Epinephrine
- C-CLAD-IL with Epinephrine: Lidocaine 2% and 1:100,000 Epinephrine
  Interventions: Procedure: C-CLAD-IL with Epinephrine
- Infiltration with Epinephrine: Lidocaine 2% and 1:100,000 Epinephrine
  Interventions: Procedure: Infiltration with Epinephrine
- Mandibular block without Epinephrine: Mepivacain HCl 3% without Epinephrine
  Interventions: Procedure: Mandibular block without Epinephrine
- Infiltration without Epinephrine: Mepivacain 3% without Epinephrine
  Interventions: Procedure: nfiltration without Epinephrine
- CCLAD-IL without Epinephrine: Mepivacain HCl 3% without Epinephrine
  Interventions: Procedure: C-CLAD-IL without Epinephrine

INTERVENTIONS:
Procedure: mandibular block with Epinephrine — Delivery of mandibular block anesthesia for dental treatment with Lidocaine HCl 2% with 1:100,000 Epineprine
  Groups: Mandibular block with Epinephrine
Procedure: C-CLAD-IL with Epinephrine — Delivery of C-CLAD-ILanesthesia for dental treatment with Lidocaine HCl 2% with 1:100,000 Epineprine
  Groups: C-CLAD-IL with Epinephrine
Procedure: Infiltration with Epinephrine — Delivery of infiltration anesthesia for dental treatment with Lidocaine HCl 2% with 1:100,000 Epineprine
  Groups: Infiltration with Epinephrine
Procedure: Mandibular block without Epinephrine — Delivery of mandibular block anesthesia for dental treatment with Mepivacaine 3% without Epineprine
  Groups: Mandibular block without Epinephrine
Procedure: C-CLAD-IL without Epinephrine — Delivery of C-CLAD-ILanesthesia for dental treatment with Mepivacaine 3% without Epineprine
  Groups: CCLAD-IL without Epinephrine
Procedure: nfiltration without Epinephrine — Delivery of infiltration anesthesia for dental treatment with Mepivacaine 3% without Epineprine
  Groups: Infiltration without Epinephrine

SUMMARY:
Incident and extent of pulse alteration during administration of various modes of local anesthesia in children during routine dental treatment. Our aims are: (1) To estimate the percent of patients who receive mandibular block , C-CLAD-IL or infiltration injections and show increase in their pulse rate during the delivery of anesthesia (in spite of negative aspiration) as result of infiltration of adrenalin into their blood vessels. (2) To estimate the extent of pulse rate alteration in correlation with the velocity or volume of local anesthesia injected. (3) To examine the correlation between increase in the pulse rate and effectiveness of anesthesia. (4) To examine the correlation between the needle gauge (27 & 30) and increase in pulse rate during mandibular block injection in spite of negative aspiration. We will recruit children that undergo routine dental treatment under local anesthesia (such as mandibular block, infiltration or C-CLAD-IL). Patients will be connected, immediately before and during the entire delivery of the local anesthetic, to pulse-oximeter that will be connected to a computer and continuously monitor pulse rate and saturation during the delivery of local anesthesia. Each aberrant event which may occur during alteration of the pulse rate such as gag reflex, coughing, or pain related disruptive behavior will be documented on the computer in real time by another person that is not the treating dentist. All types of local anesthesia delivery will be performed by the computerized-controlled local anesthesia delivery system - Single-Tooth-Anesthesia which connected to a computer and documents continuously the amount and velocity of the local anesthetic delivered to the patient. All injections will be performed by using a 29 gauge needle, except when children will be treated under general anesthesia, the injection will be performed also by 27 gauge needle. In case the pulse rate will increase to 150% of the baseline rate, or when the pulse will reach 150 beats/minute the injection will be stopped immediately. The continuation of the local anesthetic delivery will be continued in different location and only after the return of the pulse to its basic rate. A total of 100 patients will receive local anesthetic containing 1:100,000 adrenalin and 50 patients without adrenaline. Three modes of local anesthesia will be evaluated: C-CLAD-IL, infiltration and mandibular block= a total of 300 patients.

DETAILED DESCRIPTION:
Parents to children (healthy and with systemic disease ) who need local anesthesia (such as mandibular block, infiltration or C-CLAD-IL) for routine dental treatment will be asked to sign an informed consent form to participate in the study. The parents will receive explanation that the aim of the study is to evaluate the alteration of the pulse rate during delivery of different modes of local anesthetic delivery (an indirect sign for penetration of local anesthetic solution into the blood vessels). All patients will be connected, immediately before and during the entire delivery of the local anesthetic, to pulse oximeter ( pulse oximeter ,Boston, USA Nellcor N550) . The probe will be attached to the patient's finger or big toe according to patient's age. The pulse oximeter will be connected to a computer that will document continuously the pulse rate and saturation during the delivery of local anesthesia. Each aberrant event which may occur during alteration of the pulse rate such as gag reflex, coughing, or pain related disruptive behavior (crying, grimace, body movements or verbal complains-CHEOPS, attachment 1) will be documented on the computer in real time by another person that is not the treating dentist. This documentation is feasible due to a new program that was developed especially for this study. All types of local anesthesia delivery will be performed by the computerized controlled local anesthesia delivery system - Single-Tooth-Anesthesia (C-CLAD, STA, Milestone Scientific, Inc. Deerfield, IL, USA) which connected to a computer and documents continuously the amount and velocity of the local anesthetic delivered to the patient. This program was kindly provided and developed by Dr. Mark Hochman from USA, as part of the collaboration in the present study.

The local anesthesia will be performed by using Lidocaine 2% and Epinephrine 1:100,000, or Mepivacain HCl 3% without any vasoconstrictors as necessary. The use of local anesthetic without vasoconstrictor will serve as control for elevations of pulse rate which not resulted from penetration of adrenalin into the blood vessels.

When injecting mandibular block or infiltration, aspiration will be performed immediately before injecting the solution. In case a positive aspiration, the finding will be marked; the location of the needle will be changed until a negative aspiration will be received.

All injections will be performed by using a 29 gauge needle, except when children will be treated under general anesthesia, the injection will be performed also by 27 gauge needle.

In case the pulse rate will increase to 150% of the baseline rate, or when the pulse will reach 150 beats per minute the injection will be stopped immediately. The continuation of the local anesthetic delivery will be continued in different location and only after the return of the pulse to its basic rate.

When performing mandibular block injection, the lingual and buccal nerves will be anesthetized as well. The total injected volume during mandibular block delivery will be 1.8 ml. In case full anesthesia is not achieved (after waiting 5 minutes) additional injection will be performed. In any case the amount of local anesthetic injected will not exceed the amount of 4.4 mg/kg body weight.

When a participating child will be scheduled to two consecutive appointments for similar treatments, the child will receive in one appointment local anesthesia without adrenalin and in the other with adrenalin or vice versa.

Anesthesia effectiveness. The dentist will assess the effectiveness of anesthesia through the presence or absence (non-contiguous) of pain-disruptive behavior during treatment as described by Oulis et al. (6). Each single sign of discomfort (even mild) was rated as a positive presence of pain. Signs of discomfort included visual or acoustic changes, such as hand or body tension or movements, eye movements, verbal complaints, or tears. Anesthesia will be rated adequate only when the child will be completely relaxed during treatment.

Each patient will have a computerized file in which his details will be filled The name of the treating dentist Name of the patient Systemic disease Type of management: behavior management, nitrous oxide, sedation , general anesthesia Type of local anesthesia Number of tooth Type of local anesthetic solution: Lidocaine 2% and 1:100,000 Epinephrine, Mepivacaine HCl 3% without Epinephrine Gauge of the needle 30 gauge or 27 gauge Side of injection Number of positive aspiration Number of negative aspirations Type of treatment provided Effective of local anesthesia during treatment Basic pulse rate before injection Maximum pulse during injection The reason for the increasing pulse rate: gag reflex, coughing, pain, bitter test, nothing

All details will be completed before during or immediately after completing the injection.

Number of patients 100 patients for each mode of anesthesia 50 patients will receive local anesthetic containing 1:100,000 Epinephrine and 50 patients without Epinephrine Three modes of local anesthesia will be evaluated: C-CLAD-IL, infiltration and mandibular block= 300 patients Each patient will participate maximum twice in each mode of anesthesia ( once will receive local anesthetic containing 1:100,000 Epinephrine and 50 patients without Epinephrine). The type of local anesthesia solution will be selected by the dentist according to the patient's need and will not be affected by the study. Children who do not fully cooperate during treatment will be excluded from the present study.

Attachent 1: CHOPES items Item Behavior Score Definition Cry no cry 1 Child is not crying moaning 2 Child is moaning or quickly crying 2 Child is crying but the cry is gentle or whimpering scream 3 Child is in a full-lunged cry; sobbing may be scored with complaint or without complaint: Facial composed 1 Neutral facial expression grimace 2 Score only if definite negative facial expression smiling 0 Score only if definite negative facial expression Child verbal none 1 Child is not talking. other complains 1 Child complains but not about pain, e.g., I want to see my mommy," or "I am Thirsty " pain complaints 2 Child complains about pain both complaints 2 Child complains about pain and about other things, e.g., "It hurts; I want mommy" positive 0 Child makes any positive statement or talks about other things without complaint. Torso neutral 1 Body (not limbs) is at rest; torso is inactive. shifting 2 Body is in motion in a shining or serpentine tense 2 Body is arched or rigid. shivering 2 Body is shuddering or shaking involuntarily. upright 2 Child is in vertical or upright position. restrained 2 Body is restrained. Touch not touching 1 Child is not touching or grabbing at wound reach 2 Child is reaching for but not touching wound. touch 2 Child is gently touching wound or wound area. grab 2 Child is grubbing vigorously at wound. restrained 2 Child's arms are restrained. Legs neutral 1 Legs may be in any position but are relaxed included gentle swimming or serpentine- like movements. Squirming\ kicking\ drawn up 2 Definitive uneasy or restless movements in the legs and/or striking out with foot or feet.

tense 2 Legs tensed and/or pulled up tightly to body and kept there standing 2 Standing. crouching. or kneeling restrained 2 Child's legs are being held down.

ELIGIBILITY:
Inclusion Criteria:

All children that their parents signed the inform consent form and the children allow to put the pulse oximeter sensor on their finger/ear.

Exclusion Criteria:

Children that does not allow to put the pulse oximeter sensor on their finger/ear.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children undergo routine dental treatment that require local anesthetic.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Pulse rate alteration (1-90 beates) | 10 minutes, during entire delivery of local anesthesia
  increase pulse rate above 50% of the baseline rate, or when the pulse will reach 150 beats/minute the injection will be stopped immediately.